CLINICAL TRIAL: NCT02811289
Title: Pharmacological or Cold-induced Activation of Brown Adipose Tissue Metabolism
Brief Title: Pharmacological Activation of Brown Adipose Tissue Metabolism
Acronym: GB6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, André Carpentier, Tenured professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-1086
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mirabegron

ARMS (2):
- Mirabegron (Experimental): Mirbetriq (Mirabegron) (50mg) will be administered orally at time 0 to activate brown adipose tissue.
  Interventions: Drug: Mirbetriq (Mirabegron); Radiation: injection of 18FDG; Radiation: injection of 11C-acetate; Radiation: [3-3H]-glucose; Other: [U-13C]-palmitate; Other: 2H-Glycerol
- Cold exposure (Active Comparator): Cold exposure protocol using a water-conditioned cooling suit will be applied
  Interventions: Other: cold exposure; Radiation: injection of 18FDG; Radiation: injection of 11C-acetate; Radiation: [3-3H]-glucose; Other: [U-13C]-palmitate; Other: 2H-Glycerol

INTERVENTIONS:
Drug: Mirbetriq (Mirabegron) — 50mg of Mirabegron will be administered orally at time 0 in protocol A.
  Other Names: Mirabegron
  Arms: Mirabegron
Other: cold exposure — Acute cold exposure protocol using a water-conditioned cooling suit will be applied from time 120 to 300 min in protocol B
  Arms: Cold exposure
Radiation: injection of 18FDG — I.v. injection of 18-fluorodeoxyglucose (18FDG) will be performed at time 270 min, followed by 30 min dynamic PET/CT scanning
Radiation: injection of 11C-acetate — i.v. injection of 11C-acetate will be performed, followed by 20 min dynamic PET/CT scanning
Radiation: [3-3H]-glucose — i.v. administration of 1.5 uCi/min of [3-3H]-glucose
Other: [U-13C]-palmitate — i.v. administration of 0.08 umol/kg/min of [U-13C]-palmitate
Other: 2H-Glycerol — i.v. administration of 0.05 µmol/kg/min of 2H-glycerol

SUMMARY:
Lean tissue intracellular triglycerides (ICTG) accretion is an important marker of lean tissue lipotoxicity that significantly contributes to the development of type 2 diabetes (T2D). The mechanisms leading to excess exposure of lean tissues to fatty acids involve metabolic dysfunctions of adipose tissues and lean tissues themselves. Understanding the role of white and brown adipose tissue in this metabolic dysfunction is particularly important in predicting, preventing and treating T2D and many of its associated cardiovascular complications.

A recent breakthrough has been the demonstration that the acute oral administration of a β3 adrenergic agonist, mirabegron (200 mg), significantly increases BAT glucose uptake in healthy individuals. This suggests that mirabegron could be used as a pharmacological tool to selectively activate BAT metabolism as part of the mechanistic studies on BAT. It also suggests that mirabegron could be used pharmacologically for chronic activation of BAT in clinical trials to treat obesity and T2D. However, there are some outstanding issues regarding the use of mirabegron to activate BAT. First, there has been no direct comparison of the effect of acute cold vs. mirabegron on BAT metabolism. Second, there has been no demonstration of the effect of mirabegron on BAT oxidative metabolism since glucose uptake is only a surrogate of BAT energy expenditure. Third, acute administration of mirabegron led to significant increases in blood pressure and cardiac work, suggesting that it may also enhance energy expenditure in other organs in addition to BAT, thus confounding the role of BAT in energy homeostasis. Therefore, much remains to be known about the effect of mirabegron on BAT and cardiac energy metabolism before this drug can be used as a selective activator of BAT oxidative metabolism. The purpose of this study is to directly compare BAT oxidative metabolism under cold vs. β3-adrenergic agonist stimulation in lean healthy individuals. The investigator hypothesizes that the acute oral administration of a lower dose of mirabegron (50 mg) will result in an increase in BAT oxidative metabolism and whole-body energy expenditure, to a similar extent as cold exposure, without influencing the cardiovascular responses previously seen with the higher dose (200 mg).

DETAILED DESCRIPTION:
The first step of the study will be direct comparison of mirabegron (protocol A) vs. cold-induced (protocol B) BAT metabolic activation using 11C-acetate to measure BAT metabolic activity. The principle of this method is measurement of tissue fast disappearance of 11C, a marker of tissue 11CO2 production. This fast tissue 11C clearance thus gives an index of tissue oxidative metabolism. Ten healthy, non obese men will undergo two identical 5h procedures in which BAT metabolism will be stimulated with a β3-agonist (mirabegron 50mg) or using cold exposure, in random order. The investigator just received approval from Health Canada to use mirabegron as part of these metabolic investigations. In brief, baseline blood samples and indirect calorimetry will be performed between time -60 to -30 min followed by i.v. injection of 11C-acetate with 30 min dynamic PET/CT scanning at room temperature in both protocol A and B. Mirabegron will be administered orally at time 0 in protocol A whereas acute cold exposure protocol using a water-conditioned cooling suit will be applied from time 120 to 300 min in protocol B. At time 210 min (i.e. Tmax of plasma mirabegron level or 90 min after the onset of cold exposure), i.v. injection of 11C-acetate will be repeated followed by 30 min dynamic PET/CT scanning. I.v. injection of 18-fluorodeoxyglucose (18FDG) will be performed at time 270 min, followed by 30 min dynamic PET/CT scanning to determine BAT net glucose uptake and a whole-body PET/CT scan to determine BAT volume of metabolic activity and organ-specific glucose partitioning.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* normal glucose tolerance (2-hour post 75g OGTT glucose at < 7.8 mmol/l
* HbA1c < 5.8%

Exclusion Criteria:

* overt cardiovascular disease as assessed by medical history, physical exam, and abnormal ECG;
* treatment with any drug known to affect lipid or carbohydrate metabolism;
* presence of liver or renal disease, uncontrolled thyroid disorder, previous pancreatitis, bleeding disorder, or other major illness;
* smoking (>1 cigarette/day) and/or consumption of >2 alcoholic beverages per day;
* prior history or current fasting plasma cholesterol level > 7 mmol/l or fasting TG > 6 mmol/l.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
BAT net glucose uptake | 2 years
  will be assessed using i.v. injection of 18FDG with sequential dynamic PET/CT scanning.
BAT oxidative metabolism | 2 years
  will be determined using i.v. injection of 11C-acetate during dynamic PET/CT scanning
BAT volume of metabolic activity | 2 years
  will be determined using a total body CT (16 mA) followed by a PET acquisition.
whole body organ glucose partitioning | 2 years
  will be determined using a total body CT (16 mA) followed by a PET acquisition be determined using a total body CT (16 mA) followed by a PET acquisition

SECONDARY OUTCOMES:
lipolysis rate | 2 years
  will be measured using i.v. administration of [13C]-palmitate and [2H]-glycerol, using steele's non steady state equations
Glucose appearance rate | 2 years
  will be determined using [3-3H]-glucose
Energy expenditure | 2 years
  will be determined by indirect calorimetry from VO2 and VCO2 (Vmax29n, Sensormedics)
Insulin sensitivity | 2 years
  will be determined using the HOMA-IR (based on fasting insulin and glucose levels)
Insulin secretion rate | 2 years
  will be assessed using deconvolution of plasma C-peptide with standard C-peptide kinetic parameters
β-cell function | 2 years
  will be assessed by calculation of the disposition index (DI) that is insulin secretion in response to the ambient insulin sensitivity.
metabolite responses | 2 years
  will be determined using a multiplex assay system
Electrocardiogram | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: André Carpentier, M.D., Principal Investigator — Centre de recherche du CHUS
Locations (1):
- centre de recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Blondin DP, Nielsen S, Kuipers EN, Severinsen MC, Jensen VH, Miard S, Jespersen NZ, Kooijman S, Boon MR, Fortin M, Phoenix S, Frisch F, Guerin B, Turcotte EE, Haman F, Richard D, Picard F, Rensen PCN, Scheele C, Carpentier AC. Human Brown Adipocyte Thermogenesis Is Driven by beta2-AR Stimulation. Cell Metab. 2020 Aug 4;32(2):287-300.e7. doi: 10.1016/j.cmet.2020.07.005. PMID 32755608